CLINICAL TRIAL: NCT07406464
Title: The Impact of tDCS on Substrates of Emotion Processing Using fMRI in Healthy Volunteers
Brief Title: MRI-tDCS Criticism Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Collaborators: University Ghent (Other)
Responsible Party: Principal Investigator, Sara De Witte, Dr., Universitair Ziekenhuis Brussel
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: Approved by UZ Gent EC
Record Dates: First submitted 2025-11-26; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-12

CONDITIONS: Healthy Participant Study
Keywords: tDCS; Criticism; neuronavigation; DLPFC; fMRI; MRI; DNA; ASL
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active tDCS (Active Comparator): Participants receive MRI-compatible transcranial direct current stimulation (tDCS) using a NeuroConn DC-Stimulator MR. A constant current of 1.5 mA is applied for 20 minutes with the anodal electrode positioned over the left dorsolateral prefrontal cortex (DLPFC) using neuronavigation and the cathodal electrode positioned over the contralateral supra-orbital area. Stimulation is delivered while participants are in the MRI scanner.
  Interventions: Device: tDCS
- Sham tDCS (Placebo Comparator): Participants receive sham MRI-compatible transcranial direct current stimulation using a NeuroConn DC-Stimulator MR. The electrodes are positioned identically to the active condition. The current is ramped up and down during the first 30 seconds to mimic the initial sensation of stimulation, after which no current is delivered for the remainder of the 20-minute session. Stimulation is administered while participants are in the MRI scanner.
  Interventions: Device: tDCS

INTERVENTIONS:
Device: tDCS — Participants are randomized to receive either active or sham tDCS during MRI scanning. Neuroimaging and behavioral outcomes are used to assess the effects of stimulation on emotion-related brain networks.

SUMMARY:
This experimental study investigated how MRI-compatible transcranial direct current stimulation (tDCS) over the left dorsolateral prefrontal cortex (DLPFC) modulates neural and cognitive responses to social criticism in healthy volunteers.

Participants underwent two MRI sessions - one with active and one with sham stimulation - in a randomized, double-blind, cross-over design.

During stimulation, they completed resting-state and task-based fMRI scans including exposure to critical, neutral, and praising auditory comments, followed by behavioral and self-report measures of rumination, mood, and implicit self-esteem.

DETAILED DESCRIPTION:
This study aimed to examine the effects of non-invasive brain stimulation on emotional and self-referential processing. Healthy right-handed female participants completed two identical MRI sessions separated by at least 48 hours and a maximum of 2 weeks. The localization of the left dorsolateral prefrontal cortex (DLPFC) was determined during the first session. Anatomical data were first acquired using a high-resolution T1-weighted structural scan. Participants were then briefly removed from the MRI scanner to define the stimulation target using two complementary methods: (1) the standard scalp position F3 according to the 10-20 international EEG system, and (2) an individualized neuronavigation procedure targeting the mid-center of the left middle frontal gyrus (Brodmann areas 9/46) based on each participant's structural MRI. For the actual tDCS sessions, only the neuronavigation-derived DLPFC target was used for electrode placement.

In each session, participants received either active or sham MRI-compatible tDCS (1.5 mA, 20 minutes) applied over the left DLPFC with the cathode placed over the contralateral supra-orbital region. The order of stimulation (active vs. sham) was randomized and counterbalanced. The location of the DLPFC electrode placement was based During fMRI, participants completed multiple scans: a T1 structural scan, resting-state sequences (pre-, during-, and post-stimulation), resting-state sequences (pre-, during-, and post-auditory criticism task with blocks of critical, neutral, and praising comments), and an arterial spin labeling (ASL) perfusion sequence.

Self-report measures of state rumination (Momentary Ruminative Self-focus Inventory, MRSI) and mood (visual analogue scales) were collected before and after stimulation and after the criticism paradigm. An implicit self-esteem task (Implicit Relational Assessment Procedure, IRAP) followed the MRI session. Trait questionnaires and a blood sample for DNA (e.g. 5-HTTLPR) analysis were collected at baseline only.

The primary goal was to assess whether active tDCS modulates neural and behavioral markers of self-referential processing and emotional regulation compared with sham stimulation.

No serious adverse events occurred during the study. Minor sensations (tingling, mild scalp discomfort) were transient and self-limited.

ELIGIBILITY:
Inclusion Criteria:

* Female participants aged 18-35 years.
* Right-handed, healthy volunteers.
* No current or past psychiatric or neurological disorder as assessed by structured clinical interview (M.I.N.I.).
* MRI-compatible (no metal implants, pacemaker, or contraindications for MRI scanning).
* Not taking psychotropic medication.
* Fluent in Dutch.
* Provided written informed consent.

Exclusion Criteria:

* Current or past major depressive episode or any other psychiatric disorder.
* History of epilepsy or seizures in participant
* History of neurological illness or neurosurgical intervention.
* Pregnancy.
* Claustrophobia or inability to tolerate MRI environment.
* Metal implants or other MRI-incompatible devices.
* Skin lesions or dermatological conditions at electrode sites.
* Unstable medical condition.
* Use of medication that could influence brain activity or mood.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 47 (Actual)
Dates: Start 2013-07-09 (Actual); Primary Completion 2014-03-02 (Actual); Study Completion 2014-03-02 (Actual)

PRIMARY OUTCOMES:
Change in perfusion | Baseline; during tDCS; immediately post-tDCS; and immediately post-criticism paradigm (single study visit)
  Cerebral blood flow measured using arterial spin labeling (ASL) functional MRI before and after tDCS and after the criticism paradigm.
  Unit of Measure: mL/100 g/min
Neural reactivity to praise and criticism | Periprocedural
  Blood-oxygen-level dependent (BOLD) signal change during blocks of praising, neutral, and critical comments measured using task-based fMRI.
  Unit of Measure: Percent signal change (or beta values from the general linear model)
Resting-state functional connectivity within emotion-regulation networks | Baseline; immediately post-tDCS; and immediately post-criticism paradigm (single study visit)
  Functional connectivity strength between prefrontal and limbic regions measured using resting-state fMRI before, during, and after tDCS.
  Unit of Measure: Fisher-z transformed correlation coefficients

SECONDARY OUTCOMES:
Change in momentary rumination | Baseline; immediately post-tDCS; and immediately post-criticism paradigm (single study visit)
  Momentary rumination assessed using the Perseverative Thinking Questionnaire (PTQ).
  Unit of Measure: PTQ total score. A higher score means more rumination.
Implicit self-esteem (Implicit Relational Assessment Procedure, IRAP) | Baseline and post tDCS
  Implicit self-esteem assessed using the Implicit Relational Assessment Procedure (IRAP).
  Unit of Measure: D-IRAP score (reaction-time-based index): D-IRAP score (typically ranging approximately from -2 to +2)
Spatial deviation between targeting methods | Baseline (prior to any intervention)
  Euclidean distance between the dorsolateral prefrontal cortex (DLPFC) target coordinates derived from EEG 10-20 F3 positioning and MRI-based neuronavigation.
  Unit of Measure: Millimeters (mm)
Mood ratings-tension | Baseline; immediately post-tDCS; and immediately post-criticism paradigm (single study visit)
  Self-reported tension measured using a visual analogue scale (VAS) Unit of Measure: Score on a 0-10 scale. A higher score means more tensed.
Momentary mood ratings - fatigue | Baseline; immediately post-tDCS; and immediately post-criticism paradigm (single study visit)
  Self-reported fatigue measured using a visual analogue scale (VAS).
  Unit of Measure:Score on a 0-10 scale. A higher score means more fatigued.
Momentary mood ratings - vigor | Baseline; immediately post-tDCS; and immediately post-criticism paradigm (single study visit)
  Self-reported vigor measured using a visual analogue scale (VAS).
  Unit of Measure: Score on a 0-10 scale. A higher score means more vigor.
Momentary mood ratings - anger | Baseline; immediately post-tDCS; and immediately post-criticism paradigm (single study visit)
  Self-reported anger measured using a visual analogue scale (VAS).
  Unit of Measure: Score on a 0-10 scale. A higher score means more anger.
Momentary mood ratings - depressed mood | Baseline; immediately post-tDCS; and immediately post-criticism paradigm (single study visit)
  Self-reported depressed mood measured using a visual analogue scale (VAS).
  Unit of Measure: Score on a 0-10 scale. A higher score means more depressed mood.
Momentary mood ratings - cheerfulness | Baseline; immediately post-tDCS; and immediately post-criticism paradigm (single study visit)
  Self-reported cheerfulness measured using a visual analogue scale (VAS).
  Unit of Measure: Score on a 0-10 scale. A higher score means more cheerfulness.

OTHER OUTCOMES:
Serotonin transporter genotype | Baseline (prior to any intervention)
  Serotonin transporter promoter polymorphism (5-HTTLPR) determined from baseline DNA samples.
  Unit of Measure: Genotype category (e.g., LL, LS, SS)
Temperament and Character Inventory (TCI) | Baseline (prior to any intervention)
  Temperament and character traits assessed using the Temperament and Character Inventory (TCI).
  Unit of Measure: TCI-240 true/false items. Temperament traits assessed using the TCI (NS, HA, RD, P subscales) and Character traits assessed using the TCI (SD, C, ST subscales).
  TCI subscale scores (NS 0-40; HA 0-35; RD 0-24; P 0-8; SD 0-44; C 0-42; ST 0-33)
  Higher scores indicate greater expression of that trait.
Perceived criticism sensitivity | Baseline (prior to any intervention)
  Perceived criticism assessed using the Perceived Criticism Measure (PCM), a single-item rating of how critical a significant other is perceived to be.
  Unit of Measure: PCM score (range 1-10; higher scores indicate greater perceived criticism)
Trait anxiety | Baseline (prior to any intervention)
  Trait anxiety assessed using the State-Trait Anxiety Inventory - Trait version (STAI-T).
  Unit of Measure: STAI-T total score (range 20-80; higher scores indicate greater trait anxiety).
Explicit self-esteem | Baseline (prior to any intervention)
  Explicit self-esteem assessed using the Rosenberg Self-Esteem Scale (RSES).
  Unit of Measure: RSES total score (range 10-40; higher scores indicate higher self-esteem).
Psychological inflexibility | Baseline (prior to any intervention)
  Psychological inflexibility assessed using the Acceptance and Action Questionnaire-II (AAQ-II).
  Unit of Measure: AAQ-II total score (range 7-49; higher scores indicate greater psychological inflexibility)
Cognitive emotion regulation strategies | Baseline (prior to any intervention)
  Cognitive emotion regulation strategies assessed using the Cognitive Emotion Regulation Questionnaire (CERQ).
  Unit of Measure:Cognitive emotion regulation strategies assessed using the CERQ, reported as subscale scores. CERQ subscale scores each ranging 4-20. A higher score means less Cognitive emotion regulation strategies.
Trait rumination | Baseline (prior to any intervention)
  Trait rumination assessed using the Ruminative Responses Scale (RRS).
  Unit of Measure: RRS total score (range 22-88; higher scores indicate greater trait rumination).

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Gent, Ghent, Oost-Vlaanderen, Belgium

IPD SHARING:
Plan to Share IPD: No